CLINICAL TRIAL: NCT04873661
Title: Hypnosis, Meditation and Cognitive Trance on Cancer Patients: Impact on Quality of Life and Neurophysiology
Brief Title: Cognitive Trance, Hypnosis and Meditation in Oncology
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: FNRS (Télévie) (Unknown); Fondation contre le cancer (Unknown); Bial Foundation (Unknown); Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, PhD in Medical Sciences, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Trance-Onco
Record Dates: First submitted 2021-04-26; First posted 2021-05-05 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Distress, Emotional; Pain; Fatigue; Sleep Disturbance; Cognitive Impairment
Keywords: Hypnosis; Cognitive trance; Meditation; Cancer; Oncology; Quality of life; Neurophysiology; Phenomenology
MeSH Terms: conditions — Neoplasms; Pain; Fatigue; Parasomnias; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hypnosis (Experimental): In the hypnosis-based intervention, patients (in groups of approximately 10 participants) will participate in 8 weekly sessions (2 hours each) during which they will benefit from guided hypnosis exercises, and learn how to implement self-hypnosis. They will also receive a CD with hypnosis exercises for home practice. At-home practice is encouraged between sessions.
  Interventions: Behavioral: Hypnosis group intervention
- Cognitive trance (Experimental): The cognitive trance-based intervention will consist of a two-day workshop in groups of approximately 10 participants, where they will learn how to induce the cognitive trance, with the use of different sound-loops that can induce trance in untrained people in a safe way. After two weeks of home practice, participants will redo a two-day consolidation training. At-home practice is encouraged between sessions.
  Interventions: Behavioral: Cognitive trance group intervention
- Meditation (Experimental): The meditation-based intervention will consist of 8 weekly sessions (2h45 each) in groups of approximately 10 participants, as well as half a day of intensive practice between the fifth and the sixth session. Participants will learn how to implement self-compassion meditation, through practical exercises proposed during the sessions. At-home practice is encouraged between sessions.
  Interventions: Behavioral: Meditation group intervention
- Control group (No Intervention): Participants in the control group will not receive any intervention during the whole duration of the study. They will be assessed at the same times and in the same ways than the 3 experimental groups. After the study, they will have the opportunity to participe in one of the 3 interventions if they want to.

INTERVENTIONS:
Behavioral: Hypnosis group intervention — See arm description
  Arms: Hypnosis
Behavioral: Cognitive trance group intervention — See arm description
  Arms: Cognitive trance
Behavioral: Meditation group intervention — See arm description
  Arms: Meditation

SUMMARY:
Patients with cancer often suffer from a symptom cluster, including pain, fatigue, sleep difficulties, emotional distress and cognitive impairments. In oncology settings, there is a growing interest in "mind-body" intervention, to relieve them in a non-pharmacological way. Hypnosis and meditation are two modified state of consciousness shown to positively this symptom cluster. Cognitive trance is also a modified state of consciousness, but is induced by body movements and/or vocalizations. Subjective reports of experts in cognitive trance showed a modification of self, emotion regulation, pain perception, attention and concentration. However, we still need to develop studies to better characterise this particular state of consciousness and its clinical applications. Our randomized-controlled trial aims at comparing both interventions in terms of (1) benefits on cancer patients' quality of life (pain, fatigue, sleep, distress, cognitive impairments), (2) phenomenological/subjective experiences and neurophysiological correlates, and (3) mechanisms involved in patients' responsiveness, based on the biopsychosocial model of hypnosis.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* No neurological/psychiatric disorders/history of alcohol or drug abuse
* No current and regular practice of hypnosis, meditation or cognitive trance
* Diagnosis of cancer (all localisations accepted except brain tumours to avoid any effect on EEG data and cognitive impairments)
* Active treatments (surgery, chemotherapy, radiotherapy) finished for less than a year.
* Score of at least 4/10 for one of these four symptoms at baseline: pain, fatigue, sleep difficulties, emotional distress.

Exclusion Criteria:

* < 18 year old
* No cancer diagnosis
* Neurological or psychiatric disorder
* Brain tumour ou other tumour with brain metastases
* Active treatments still ongoing or finished for more than a year
* No baseline symptom at 4/10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Fatigue | Assessed before the intervention (T0), immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Assessed with a questionnaire (Multidimensional Fatigue Inventory; MFI-20)
Change in Pain | Assessed before the intervention (T0), immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Assessed with a visual analogue scale (VAS) (score range from 0 to 10/10, a higher score indicating a higher pain)
Change in Sleep difficulties | Assessed before the intervention (T0), immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Assessed with a questionnaire (Insomnia Severity Index; ISI). Score range from 0 to 28, with a higher score indicating higher sleep difficulties.
Change in Emotional distress | Assessed before the intervention (T0), immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Assessed with a questionnaire (Hospital Anxiety and Depression Scale; HADS). Score range from 0 to 42, with a higher score indicating higher emotional distress
Change in Perceived cognitive difficulties | Assessed before the intervention (T0), immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Assessed with a questionnaire (FACT-Cog), investigation 4 dimensions (perceived cognitive impairments, score range 0-72, higher score indicating less impairments ; impact of cognitive impairments on quality of life, score range 0-16, with higher scoe indicating less impact ; Comments from others, score range 0-16 with higher score indicating less comments ; perceived cognitive abilities, score range 0-28, with higher score indicating more cognitive abilities)

SECONDARY OUTCOMES:
Change in Psychological flexibility | Assessed before the intervention (T0), immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Assessed with a questionnaire (Multidimensional Psychological Flexibility Inventory; MPFI-24). Score range from 0 to 6 for each dimension (psychological flexibility and psychological inflexibility), with higher score indicating higher flexibility or inflexibility according to the dimension assessed.
Change in Mental Adjustment to Cancer | Assessed before the intervention (T0), immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Assessed with a questionnaire (Mental adjustment to cancer; MAC). 2 summary scores (Summary positive adjustment, score range from 17 to 68, with higher score indicating higher positive adjustmen ; Summary Negative Adjustment, score ranging from 16 to 64, with higher score indicating highr negative adjustment)
Change in Emotion regulation | Assessed before the intervention (T0), immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Assessed with a questionnaire (Cognitive Emotion Regulation Questionnaire; CERQ). 2 summary scores (adpative regulation, score ranging from 20 to 100, with higher score indicating higher adaptive regulation ; non-adaptive regulation, score ranging 12-60, with higher score indicating higher non-adaptive regulation)
Change in Empowerment | Assessed before the intervention (T0), immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Assessed with a questionnaire composed of 7 VAS (score from 0 to 10/10, with higher score indicating higher empowerment), based on the Health Education Impact Questionnaire (heiQ)
Personnality characteristics | Assessed before the intervention (T0)
  Assessed with a questionnaire (Big Five Short Form; BFI-10). 5 scales (extraversion, agreeableness, conscientiousness, neuroticism, openness to experience) with score range 1-5, with higher score indicating a stronger presence of this personality trait.
Fantasy Proneness (imaginative experiences) | Assessed before the intervention (T0)
  Assessed with a questionnaire designed by our team investigating the previous imaginative experiences of the participant. 25 true/false items. Total score ranging from 0 to 25, with higher score indicating higher level of fantasy proneness.
Expectations and motivation to participate in the chosen intervention | Assessed before the intervention (T0)
  Assessed with 2 VAS (score range from 0 to 10/10, with higher score indicating higher motivation and higher expectations)
Personal definition of hypnosis/cognitive trance/meditation | Assessed before the intervention (T0)
  Free text written by the participant
Change in the characteristics of a free recall of an intense hypnosis/cognitive trance/meditation episode (or an intense autobiographical episode for the participants in the control group) | Assessed immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Free text written by the participant
Change in Characteristics of the intense memory described above | Assessed immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Assessed with a questionnaire (Memory Characteristics Questionnaire; MCQ). Score range from 8 to 104, with higher score indicating higher degree of details about the memory.
Change in Mystical characteristics of the intense memory described above | Assessed immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Assessed with a questionnaire (Revised Mystical Characteristics Questionnaire; MEQ-30). 4 scales (mystical, score range 0-75, with higher score indicating a more mystical experience ; Positive mood, score range 0-30, with higher score indicating more positive mood during the episode ; Transcendence of time and space, score range 0-30, with higher score indicating stronger trenscendence ; Ineffability, score range 0-15, with higher score indicating higher ineffability)
Change in presence during the intense memory described above | Assessed immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Assessed with a questionnaire designed by our team to assess the feeling of presence in the imaginative environment linked to the intense memory reported (hypnosis, trance, meditation or personal memory). 2 scales (Presence in the suggested environment and Interaction with others, score range for each dimension 6-42, with higher score indicating higer presence/interaction).
Change in the quality of the relationship with the therapist who animated the group sessions | Assessed immediately after the intervention (T1), and at 3- and 12-month follow-up (T3 and T4)
  Assessed with a VAS (score range from 0 to 10/10, with higher score indicating better relationship quality).
Change in cerebral activity | Resting state : Assessed before the intervention (T0), immediately after the intervention (T1), and at 12-month follow-up (T4). During hypnosis, trance or meditation : T1, T4.
  Assessed with an electroencephalogram (EEG), during resting state and during hypnosis, trance or meditation, according to the chosen intervention. During the EEG, we will also measure the heart rate (with an electrocardiogram), the body temperature, the body movements (with an electromyogram) and the respiration amplitude.
Change in heart rate | Resting state : Assessed before the intervention (T0), immediately after the intervention (T1), and at 12-month follow-up (T4). During hypnosis, trance or meditation : T1, T4.
  During the EEG, heart rate will be measured (with an electrocardiogram).
Change in body movements | Resting state : Assessed before the intervention (T0), immediately after the intervention (T1), and at 12-month follow-up (T4). During hypnosis, trance or meditation : T1, T4.
  During the EEG, body movements will be measured (with an electromyogram).
Change in body temperature | Resting state : Assessed before the intervention (T0), immediately after the intervention (T1), and at 12-month follow-up (T4). During hypnosis, trance or meditation : T1, T4.
  During the EEG, body temperature will be measured (with a dedicated electrode put on the chest).
Change in respiration | Resting state : Assessed before the intervention (T0), immediately after the intervention (T1), and at 12-month follow-up (T4). During hypnosis, trance or meditation : T1, T4.
  During the EEG, respiration (amplitude, effort) will be measured (with a dedicated belts put on the torso)

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Gosseries, PhD, Principal Investigator — ULiège
Locations (1):
- University of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baussard L, Ernst M, Diep A, Jerusalem G, Vanhaudenhuyse A, Marie N, Bragard I, Faymonville ME, Gosseries O, Gregoire C. Network Analyses Applied to the Dimensions of Cancer-Related Fatigue in Women With Breast Cancer. Cancer Med. 2024 Oct;13(19):e70268. doi: 10.1002/cam4.70268. PMID 39387227
- [Derived] Gregoire C, Marie N, Sombrun C, Faymonville ME, Kotsou I, van Nitsen V, de Ribaucourt S, Jerusalem G, Laureys S, Vanhaudenhuyse A, Gosseries O. Hypnosis, Meditation, and Self-Induced Cognitive Trance to Improve Post-treatment Oncological Patients' Quality of Life: Study Protocol. Front Psychol. 2022 Feb 10;13:807741. doi: 10.3389/fpsyg.2022.807741. eCollection 2022. PMID 35222195